CLINICAL TRIAL: NCT04271176
Title: Liver Echinococcosis; Jaundice as Initial Presentation, Short and Long Term Results of Surgical Treatment
Brief Title: Jaundice as Initial Presentation of Liver Hydatidosis (ICTEHIDA)
Acronym: ICTEHIDA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Universidad de Extremadura (Other)
Collaborators: Complejo Hospitalario Universitario de Badajoz (Other)
Responsible Party: Principal Investigator, Gerardo Blanco-Fernández, Chief of Department, Universidad de Extremadura
Other Study IDs: UE-CHUB 002-2020
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Hepatic Echinococcosis; Jaundice
Keywords: Jaundice; Echinococcosis; Liver; Surgical treatment
MeSH Terms: conditions — Echinococcosis, Hepatic; Jaundice; Echinococcosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to evaluate patients with hepatic hydatidosis whose symptom at diagnosis was obstructive jaundice. As well as analyzing, the rate of performing preoperative ERCP, the results after surgery and morbidity

DETAILED DESCRIPTION:
Retrospective study of patients operated on for liver hydatidosis and whose initial symptom was obstructive jaundice Study period: January 2006 to September 2018

The preoperative diagnosis was based on abdominal ultrasound (US), CT scan or magnetic nuclear resonance

Surgical technique Precautions are taken to avoid the spillage of the parasite in the abdominal cavity. The peritoneal cavity is liberally protected with scolicidal agents. All patients have intraoperative ultrasound. Ultrasound is performed to locate the presence of any cysts which might not be seen by the preoperative imaging. Intraoperative ultrasound is also used to find out the relation of the cyst to the big vessels. Depending on the intraoperative findings, the location and size of the cyst will be considered the type of surgery to be performed. Radical surgery (closed and open total cystopericystectomy, or liver resection) or conservative surgery (partial cystopericystectomy, removal of the vesicles with external or internal drainage). When the cyst affects a total lobe and / or the main pedicles, a hepatectomy is performed.

The demographic data of the patients will be taken from their clinical histories. It included age, sex, medical history of hidatidosis, clinical findings, laboratory data, radiological findings, endoscopic treatment, surgical treatment.

The investigators will analyze postoperative mortality and morbidity. Complications' ranking according to the Clavien-Dindo score, 'severe complication' is defined as greater or equal to IIIa

Follow-up The follow-up of these patients will be performed with ultrasound or CT and hydatid serology. The minimum follow-up of the patients is six months. Relapse is defined as the appearance of new active liver cysts after the patient had undergone surgery.

ELIGIBILITY:
Inclusion Criteria:

* Hepatic Hydatidosis with obstructive jaundice surgically treated

Exclusion Criteria:

* Patients with conservative treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients operated on hydatidic cyst, any surgical option
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2009-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Morbidity | 90 days
  Postoperative morbidity after surgical treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Extremadura- Facultad de Medicina, Badajoz, Spain